CLINICAL TRIAL: NCT01741571
Title: Randomized Controlled Trial of Endobronchial Ultrasound Guided Fine Needle Aspiration Techniques
Brief Title: Trial of Endobronchial Ultrasound Guided Fine Needle Aspiration Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Hassan Chami, Assistant Professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: AmericanUBMC
Record Dates: First submitted 2012-11-27; First posted 2012-12-05 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Suction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EBUS guided FNA with suction (Active Comparator): Device/procedure: lymph node tissue collection using fine needle aspiration with suction applied.
  Four fine needle aspirations will be taken sequentially from each lymph node. Two with suction and two without suction applied.
  Interventions: Device: EBUS guided FNA with and without suction
- EBUS guided FNA without suction (Experimental): Device/procedure: lymph node tissue collection using fine needle aspiration without suction applied.
  Four fine needle aspirations will be taken sequentially from each lymph node. Two with suction and two without suction applied.
  Interventions: Device: EBUS guided FNA with and without suction

INTERVENTIONS:
Device: EBUS guided FNA with and without suction — Device/procedure: lymph node tissue collection using needle with and without suction applied.
  Four fine needle aspirations will be taken from each lymph node. Two with suction and two without suction applied.

SUMMARY:
Endobronchial ultrasound-guided transbronchial fine needle aspiration (EBUS-TBNA) techniques have not been well studied. The investigators will conduct a randomized study comparing the diagnostic yield and specimen quality of EBUS-FNA performed with and without suction applied.

DETAILED DESCRIPTION:
Consecutive patients with suspected malignant peribronchial masses or lymph nodes undergoing endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) will be enrolled. All participants will have 4 needle aspirations of each targeted peribronchial lesion. Two needle aspirations will be performed while applying suction and 2 needle aspirations will be performed without applying suction in random order. The investigators will compare the diagnostic yield and the quality of the specimens obtained using the two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Adult undergoing EBUS at AUBMC for suspected malignancy

Exclusion Criteria:

* Coagulopathy
* The lesion cannot be sampled because of intervening tumor or blood vessels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-12; Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of each needle aspiration technique for diagnosis of malignancy | Diagnosis of malignancy will be ascertained after 6 month clinical follow up
  A pathologist blinded to the needle aspiration technique will review the specimen obtained from each needle aspiration and will assess for presence of malignant cells.
  The sensitivity for diagnosing malignancy will be calculated and compared for the two needle aspiration technique.
Diagnostic accuracy of each needle aspiration technique for diagnosis of malignancy | Diagnosis of malignancy will be ascertained after 6 month clinical follow up
  A pathologist blinded to the needle aspiration technique will review the specimen obtained from each needle aspiration and will assess for presence of malignant cells.
  The diagnostic accuracy for diagnosing malignancy will be assessed and compared for the two needle aspiration technique.

SECONDARY OUTCOMES:
Adequacy of the needle aspiration sample | Adequacy will be assessed within 1 week from procedure
  A pathologist blinded to the needle aspiration technique will review the specimen obtained from each needle aspiration and will assess for adequacy (presence of malignant cells, granuloma or lymphocytes) The number of adequate samples will be compared for the two techniques.
Negative predicted value of each needle aspiration technique for diagnosis of malignancy | Diagnosis of malignancy will be ascertained after 6 month of clinical follow up
  A pathologist blinded to the needle aspiration technique will review the specimen obtained from each needle aspiration and will assess for presence of malignant cells.
  The negative predictive value for lack of malignant cells will be calculated and compared for the two needle aspiration techniques.
Specificity of each needle aspiration technique for diagnosis of malignancy | Diagnosis of malignancy will be ascertained after 6 month clinical follow up
  A pathologist blinded to the needle aspiration technique will review the specimen obtained from each needle aspiration and will assess for presence of malignant cells.
  The specificity for diagnosing malignant cells will be calculated and compared for the two needle aspiration techniques.
Positive predicted value of each needle aspiration technique for diagnosis of malignancy | Diagnosis of Malignancy will be ascertained after 6 month of clinical follow up
  A pathologist blinded to the needle aspiration technique will review the specimen obtained from each needle aspiration and will assess for presence of malignant cells.
  The positive predictive value for presence of malignant cells will be calculated and compared for the two needle aspiration techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Chami, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon